CLINICAL TRIAL: NCT00743496
Title: A Phase I Trial Of The Humanized Anti-GD2 Antibody (HU14.18K322A) In Children And Adolescents With Neuroblastoma, Osteosarcoma, Ewing Sarcoma and Melanoma
Brief Title: A Phase I Trial Of The Humanized Anti-GD2 Antibody In Children And Adolescents With Neuroblastoma, Osteosarcoma, Ewing Sarcoma and Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Evan T.J. Dunbar Neuroblastoma Foundation (Other); Duke University (Other); University of Wisconsin, Madison (Other); University Children's Hospital Tuebingen (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJGD2; ED FDN (Other: Evan Dunbar Neuroblastoma Foundation); NCI-2011-01150 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Neuroblastoma; Melanoma; Osteosarcoma; Ewing Sarcoma
MeSH Terms: conditions — Neuroblastoma; Melanoma; Osteosarcoma; Sarcoma, Ewing | interventions — humanized 3F8 anti-GD2 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Participants who consent to the study will receive Anti-GD2 antibody.
  Interventions: Biological: Anti-GD2 antibody

INTERVENTIONS:
Biological: Anti-GD2 antibody — Anti-GD2 antibody

SUMMARY:
Relapsed and/or refractory neuroblastoma, osteosarcoma, Ewing sarcoma and melanoma are considered difficult to treat and cure. For this study we are testing the use of a new experimental (investigational) antibody called hu14.18K322A. GD2 is expressed on the surface of most of these tumor types.

Two schedules of hu14.18K322A antibody will be evaluated in this study, (1) daily for four consecutive days schedule every 28 days and (2) once weekly for 4 weeks schedule every 28 days. Approximately 25-40 participants will be required to define the maximum tolerated dose for each schedule. Participants will continue on treatment for a maximum of 4 to 8 courses or until one or more of the criteria for off-treatment are met.

DETAILED DESCRIPTION:
SJGD2 is a Phase I dose finding study. The primary purpose of this phase I study is to determine the maximum tolerated dose (MTD) and dose-limiting toxicity of the humanized monoclonal anti-GD2 antibody, hu14.18K322A, in research participants with refractory or relapsed neuroblastoma or melanoma (Parts A and B) or osteosarcoma or Ewing sarcoma (Part C).

Initially, in Part A, one research participant will be treated at the lowest dose level of hu14.18K322A antibody [2 mg/m^2 daily for 4 consecutive days every 28 days (1 course)], and if no toxicity is observed then the next participant will be treated at the next dose level. This is continued until the first instance of biological activity (in the form of grade 2 side effects) is observed and from that point on a traditional phase I study design will be followed. A maximum of 4 courses may be given.

Part B: Hu14.18K322A antibody will be administered intravenously (IV) at a starting dose of 50 mg/m^2/dose weekly for 4 doses per course. One course is considered 28 days. A maximum of 8 courses may be given.

Part C: Hu14.18K322A antibody will be administered to 6 patients each with refractory/recurrent osteosarcoma at a maximum tolerated dose (MTD) of 60 mg/m^2 daily for 4 consecutive days every 28 days (Part C1). A cohort of patients with refractory/recurrent osteosarcoma or Ewing sarcoma will also be administered hu14.18K322A antibody at starting dose of 40 mg/m^2/dose weekly for 4 doses per course (Part C2). Participants will continue on treatment for a maximum of 8 courses.

Secondary objectives include:

1. Estimate the response rate, within the confines of a phase I study, to the humanized anti-GD2 antibody, hu14.18K322A.
2. Evaluate the pharmacokinetics of hu14.18K322A.
3. Examine whether or not human anti-human antibodies (HAHA) develop in participants receiving hu14.18K322A.
4. Assess the tolerability of the hu14.18K322A at the MTD of the daily x4 and the weekly dosing in patients with refractory or recurrent osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Part A: Recurrent or refractory neuroblastoma or melanoma.
  * Part B: Recurrent or refractory neuroblastoma or melanoma.
  * Part C: Recurrent or refractory osteosarcoma and Ewing sarcoma.
* Age: ≤ 21 years of age at the time of enrollment (i.e. participants are eligible until they reach their 22nd birthday).
* Does not have a clinically significant neurologic deficit or objective peripheral neuropathy (greater than or equal to grade 2). Peripheral (sensory or motor) neuropathy related to limb sparing procedure or amputation is allowed.
* Life expectancy: at least 8 weeks.
* Organ Function: Must have adequate organ and marrow function
* Performance status: Karnofsky ≥ 50 for > 10 years of age; Lansky ≥ 50 for children < 10 years of age.
* Prior Therapy: Patient must have fully recovered from the acute toxic effects of all prior therapy prior to enrolling on study.

  * Myelosuppressive Chemotherapy: Must not have received myelosuppressive therapy within 2 weeks prior to study entry (4 weeks if nitrosurea).
  * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with biologic agent, including retinoic acid. Participants receiving IVIG are eligible; however, participant must not receive IVIG during the 4 days of antibody infusion.
  * Radiation therapy: At least 2 weeks since prior local radiation therapy at the time of study entry.
  * Growth factors: Must not have received hematopoietic growth factors (G-CSF, GM-CSF) for at least 1 week prior to study entry.
  * Investigational agent: Must not have received investigational agent within 14 days of study entry.
  * Immune therapy: Must not have received immunosuppressive (including glucocorticoids), immunostimulatory or any immunomodulatory treatment within 2 weeks of study entry. Steroid containing inhalers, steroid replacement for adrenal insufficiency and steroid premedication for prevention of transfusion or imaging contrast agent-related allergic reaction will be permitted.
* Patients may have had prior CNS metastasis providing: CNS disease has been previously treated and CNS disease has been clinically stable for 4 weeks prior to study entry (assessment must be made by CT or MRI).
* Written informed consent following institutional and federal guidelines.

Exclusion Criteria:

* Prior monoclonal antibody: Participants having received in vivo monoclonal antibodies for biologic therapy or for tumor imaging are eligible provided they did not experience a severe allergic reaction with the antibody.
* Pregnancy or Breast Feeding: Study participants who are pregnant are not eligible for this study. Pregnancy tests must be obtained in girls who are > 10 years of age or post-menarchal within 7 days prior to study enrollment. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during participation in the trial. Breast feeding should be discontinued if a mother wishes to participate in this study.
* Allergy: known hypersensitivity to other recombinant human antibodies.
* An uncontrolled infection.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10-08 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-18 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose and dose-limiting toxicity of the humanized monoclonal anti-GD2 antibody, hu14.18K322A, in research participants with neuroblastoma, osteosarcoma, Ewing sarcoma and melanoma. | within 12 months of the start of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bishop, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Goldberg JL, Navid F, Hank JA, Erbe AK, Santana V, Gan J, de Bie F, Javaid AM, Hoefges A, Merdler M, Carmichael L, Kim K, Bishop MW, Meager MM, Gillies SD, Pandey JP, Sondel PM. Pre-existing antitherapeutic antibodies against the Fc region of the hu14.18K322A mAb are associated with outcome in patients with relapsed neuroblastoma. J Immunother Cancer. 2020 Mar;8(1):e000590. doi: 10.1136/jitc-2020-000590. PMID 32169872
- [Derived] Navid F, Sondel PM, Barfield R, Shulkin BL, Kaufman RA, Allay JA, Gan J, Hutson P, Seo S, Kim K, Goldberg J, Hank JA, Billups CA, Wu J, Furman WL, McGregor LM, Otto M, Gillies SD, Handgretinger R, Santana VM. Phase I trial of a novel anti-GD2 monoclonal antibody, Hu14.18K322A, designed to decrease toxicity in children with refractory or recurrent neuroblastoma. J Clin Oncol. 2014 May 10;32(14):1445-52. doi: 10.1200/JCO.2013.50.4423. Epub 2014 Apr 7. PMID 24711551
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols